CLINICAL TRIAL: NCT06360588
Title: MATCH Treatment Subprotocol Z1G: Phase II Study of Copanlisib in Patients With Tumors With PTEN Loss by IHC and Any PTEN Sequencing Result
Brief Title: Testing Copanlisib as Potentially Targeting Treatment in Cancers With PTEN Loss (MATCH - Subprotocol Z1G)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2024-01141; NCI-2024-01141 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); EAY131-Z1G (Other: ECOG-ACRIN Cancer Research Group); EAY131-Z1G (Other: CTEP); U10CA180820 (NIH)
Record Dates: First submitted 2024-04-10; First posted 2024-04-11 (Actual); Results first posted 2025-04-16 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Malignant Solid Neoplasm
MeSH Terms: interventions — Biopsy; Specimen Handling; copanlisib; X-Rays

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Subprotocol Z1G (PTEN loss) (Experimental): Patients receive copanlisib IV at a dose of 60 mg over 1 hour on day 18 and 15 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo tumor biopsy on study and radiologic evaluation and blood sample collection throughout the study.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Drug: Copanlisib; Procedure: Radiologic Examination

INTERVENTIONS:
Procedure: Biopsy Procedure — Undergo tumor biopsy
  Other Names: Biopsy; BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Drug: Copanlisib — Given IV
  Other Names: BAY 80 6946; BAY 80-6946; BAY 806946; BAY-80-6946; BAY806946; PI3K Inhibitor BAY 80-6946
Procedure: Radiologic Examination — Undergo radiologic evaluation
  Other Names: Radiologic Evaluation; Radiologic Exam

SUMMARY:
The phase II MATCH treatment trial tests how well copanlisib works to treat patients with cancer with PTEN loss. Copanlisib may stop the growth of tumor cells and may kill them by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the proportion of patients with objective response (OR) to targeted study agent(s) in patients with advanced refractory cancers/lymphomas/multiple myeloma.

SECONDARY OBJECTIVES:

I. To evaluate the proportion of patients alive and progression free at 6 months of treatment with targeted study agent in patients with advanced refractory cancers/lymphomas/multiple myeloma.

II. To evaluate time until death or disease progression. III. To identify potential predictive biomarkers beyond the genomic alteration by which treatment is assigned or resistance mechanisms using additional genomic, ribonucleic acid (RNA), protein and imaging-based assessment platforms.

IV. To assess whether radiomic phenotypes obtained from pre-treatment imaging and changes from pre- through post-therapy imaging can predict objective response and progression free survival and to evaluate the association between pre-treatment radiomic phenotypes and targeted gene mutation patterns of tumor biopsy specimens.

OUTLINE:

Patients receive copanlisib intravenously (IV) at a dose of 60 mg over 1 hour on day 18 and 15 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo tumor biopsy on study and radiologic evaluation and blood sample collection throughout the study.

After completion of study treatment, patients are followed up every 3 months for 2 years and then every 6 months for 1 year.

THE MATCH SCREENING TRIAL:

Please see NCT02465060 for information on the MATCH Screening Protocol and applicable documents.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have met applicable eligibility criteria in the Master MATCH Protocol EAY131/ NCI-2015-00054 prior to registration to treatment subprotocol
* Patients must fulfill all eligibility criteria outlined in Section 3.1 of MATCH Master Protocol (excluding Section 3.1.6) at the time of registration to treatment step (Step 1, 3, 5, 7)
* Patients must have complete loss of cytoplasmic and nuclear PTEN by immunohistochemistry (ICH) as determined via the MATCH Master Protocol and described in Appendix I. Patients can have any PTEN mutation or deletion status, but MUST have PTEN loss by IHC

  * NOTE: For patients entering the study, all patients must have PTEN IHC performed as described in the MATCH Master Protocol. This includes patients entering the study via the outside assay process
* Patients must not have co-existing aberrations in the MAPK or PI3K/MTOR pathways as determined by the MATCH screening assessment in NRAS, HRAS, KRAS, BRAF, PIK3CA, AKT or mTOR
* Patients must have an electrocardiogram (ECG) within 8 weeks prior to treatment assignment and must have no clinically important abnormalities in rhythm, conduction or morphology of resting ECG (e.g. complete left bundle branch block, third degree heart block)
* Patients must not have known hypersensitivity to copanlisib or compounds of similar chemical or biologic composition
* Patients must not have had prior treatment with copanlisib or other PI3K inhibitors, AKT inhibitors or mTOR inhibitors
* Patients must not be on strong inhibitors or inducers of CYP3A4 within two weeks prior to start of study treatment and for the duration of study treatment
* Patients should stop using herbal medications at least 7 days prior to the first dose of copanlisib. Herbal medications include, but are not limited to: St. John's Wort, Kava, ephedra, gingko biloba, dehydroepiandrosterone (DHEA), yohimbe, saw palmetto, black cohosh and ginseng
* Patients with type I or II diabetes mellitus must have a hemoglobulin (Hb) A1c ≤ 8.5% within 28 days from registration
* Patients must not have uncontrolled hypertension defined as systolic blood pressure (SBP) greater than 160 mmHg or diastolic blood pressure (BP) greater than 100 mmHg or use of more than 2 anti-hypertensive medications
* Patients must not have HER2 positive (3+ by IHC or fluorescence in situ hybridization [FISH] ratio ≥ 2) breast cancer
* Patients must not have indolent NHL (Non-Hodgkin's Lymphoma) or DLBCL (diffuse large B cell lymphoma) because other studies are ongoing with this agent in this group patients
* Patients must not be on anti-arrhythmic therapy other than digoxin or beta-blockers
* Absolute neutrophil count (ANC) ≥ 1.5 x 10^9 /L
* Platelets ≥ 100x10^9 /L
* Hemoglobulin (Hgb) > 9 g/dl
* Total serum bilirubin < 2.0 mg/dL
* Aspartate aminotransferase (ALT) and Alanine aminotransferase (AST) < 2.5 x upper limit of normal (ULN) (< 5 x ULN in patients with liver metastases)
* Serum creatinine < 1.5 x ULN
* Patients with non-healing wound, ulcer, or bone fracture are not eligible
* Patients with history of or current interstitial pneumonitis are not eligible. NOTE: For solid tumors, CMV PCR can be obtained at the discretion of treating physician or local institutional guidelines
* Patients must agree not to conceive or father children by agreeing to use contraception while receiving study treatment and for 1 month after the last dose of copanlisib

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2018-10-08 (Actual); Primary Completion 2023-01-05 (Actual); Study Completion 2025-12-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Jordi Rodon Ahnert, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- ECOG-ACRIN Cancer Research Group, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subprotocol Z1G was activated on June 20, 2018. Twenty-two patients were enrolled between October 2018 and September 2021. All patients were enrolled through the outside laboratory.
Pre-assignment Details: The PTEN loss status was determined by a CLIA-approved assay performed in NCI-MATCH approved laboratory for all patients in this arm. Twenty-one out of the 22 outside lab patients had their samples centrally confirmed.
Period: Overall Study
Arm/Group | Subprotocol Z1G (PTEN Loss)
Started | 22
Started Protocol Therapy | 22
Eligible and Treated | 21
Eligible, Treated and Mutation Status Confirmed (Primary efficacy analysis set) | 20
Completed | 0
Not Completed | 22
Not completed — Adverse Event | 3
Not completed — Death | 2
Not completed — Disease Progression | 14
Not completed — Withdrawal by Subject | 1
Not completed — Lack of Efficacy | 1
Not completed — Ineligible | 1

BASELINE CHARACTERISTICS:
Population: Patients who were eligible, started protocol therapy, and had mutation status confirmed at the analysis time were the analyzable patients
Arm/Group | Subprotocol Z1G (PTEN Loss)
Number analyzed (Participants) | 20
Age, Continuous [Median (Full Range); unit: years] | 62 [29 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 17
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 16
  More than one race | 1
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: ORR is defined as the percentage of patients whose tumors have a complete or partial response to treatment among analyzable patients. Objective response is defined consistent with Response Evaluation Criteria in Solid Tumors version 1.1, the Cheson (2014) criteria for lymphoma patients, and the Response Assessment in Neuro-Oncology criteria for glioblastoma patients. Details about how to define complete response and partial response can be found in the master protocol. 90% two-sided binomial exact confidence interval is calculated for ORR.
Time Frame: Tumor assessments occurred at baseline, then every 2 cycles for the first 26 cycles and every 3 cycles thereafter until disease progression, up to 3 years post registration
Population: Eligible, treated and mutation status confirmed
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Subprotocol Z1G (PTEN Loss)
Number analyzed (Participants) | 20
percentage of participants | 0 [0 to 13.9]

2. Secondary Outcome: 6-month Progression-free Survival (PFS) Rate
Description: Progression free survival is defined as time from treatment start date to date of progression or death from any cause, whichever occurs first. Disease progression was evaluated using the Response Evaluation Criteria in Solid Tumors version 1.1, the Cheson (2014) criteria for lymphoma patients, and the Response Assessment in Neuro-Oncology criteria for glioblastoma patients. Please refer to the protocol for detailed definitions of disease progression. 6 month PFS rate was estimated using the Kaplan-Meier method, which can provide a point estimate for any specific time point.
Time Frame: Assessed at baseline, then every 2 cycles for the first 26 cycles, and every 3 cycles thereafter until disease progression, up to 3 years post registration, from which 6-month PFS rate is determined
Population: Eligible, treated and mutation status confirmed
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Subprotocol Z1G (PTEN Loss)
Number analyzed (Participants) | 20
percentage of participants | 17.5 [6.0 to 34.0]

3. Secondary Outcome: Progression Free Survival
Description: PFS was defined as time from treatment start date to date of disease progression or death from any causes, whichever occurred first. Median PFS was estimated using the Kaplan-Meier method. Disease progression was evaluated using the Response Evaluation Criteria in Solid Tumors version 1.1, the Cheson (2014) criteria for lymphoma patients, and the Response Assessment in Neuro-Oncology criteria for glioblastoma patients. Please refer to the protocol for detailed definitions of disease progression.
Time Frame: Assessed at baseline, then every 2 cycles for the first 26 cycles and every 3 cycles thereafter until disease progression, up to 3 years post registration
Population: Eligible, treated and mutation status confirmed
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Subprotocol Z1G (PTEN Loss)
Number analyzed (Participants) | 20
months | 1.8 [1.4 to 3.9]

ADVERSE EVENTS:
Time Frame: Assessed every 28 days while on treatment and for 30 days after the end of treatment, up to 3 years post registration.
Description: All patients enrolled were included in the all-cause mortality analysis. Twenty-two patients were included in the toxicity analysis.
Arm/Group | Subprotocol Z1G (PTEN Loss)
All-Cause Mortality (participants affected / at risk) | 16/22
Serious Adverse Events (participants affected / at risk) | 7/22
Other Adverse Events (participants affected / at risk) | 13/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Subprotocol Z1G (PTEN Loss) (N=22)
Lymphocyte count decreased (Investigations) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Hypertension (Vascular disorders) | 2
Thromboembolic event (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Subprotocol Z1G (PTEN Loss) (N=22)
Anemia (Blood and lymphatic system disorders) | 3
Fatigue (General disorders) | 7
Diarrhea (Gastrointestinal disorders) | 4
Dyspepsia (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 8
Vomiting (Gastrointestinal disorders) | 3
Lymphocyte count decreased (Investigations) | 3
Anorexia (Metabolism and nutrition disorders) | 4
Hyperglycemia (Metabolism and nutrition disorders) | 6
Hypertension (Vascular disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2021-07-16): https://cdn.clinicaltrials.gov/large-docs/88/NCT06360588/Prot_000.pdf
  • Informed Consent Form (2021-07-16): https://cdn.clinicaltrials.gov/large-docs/88/NCT06360588/ICF_001.pdf